CLINICAL TRIAL: NCT06553573
Title: Postoperative Analgesic Efficacy Comparison of a Combination of Superficial Parasternal Block (PSB) and Recto-intercostal Fascial Plane Block (RİFPB) Versus a Combination of Erector Spinae Plane Block (ESPB) and Superficial Parasternal Block (PSB) in Patients Undergoing Cardiac Surgery With Sternotomy.
Brief Title: Comparison of PSB and RIFPB Combination With PSB and ESPB Combination in Cardiac Surgery With Sternotomy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cumhuriyet University (Other)
Responsible Party: Principal Investigator, Oguz Gundogdu, Associate Professor, Cumhuriyet University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: PSB and RİFPB vs PSB and ESPB
Record Dates: First submitted 2024-08-12; First posted 2024-08-14 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-08

CONDITIONS: Post Operative Pain
Keywords: sternotomy; cardiac surgery; parasternal block; recto-intercostal fascial plane block; erector spinae plane block; regional anesthesia; postoperative pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Parasternal Block and Recto-İntercostal Fascial Plane Block (Active Comparator): Before surgery, patients will receive a combination of bilateral PSB and RIFPB with 0.25% bupivacaine (total volume 60 ml) for postoperative pain control.
  Interventions: Other: Parasternal Block and Recto-İntercostal Fascial Plane Block
- Parasternal Block and Erector Spinae Plane Block (Active Comparator): Before surgery, patients will be given 0.25% bupivacaine (total volume 60 ml) with a combination of bilateral PSB and ESPB for postoperative pain control.
  Interventions: Other: Parasternal Block and Erector Spinae Plane Block

INTERVENTIONS:
Other: Parasternal Block and Recto-İntercostal Fascial Plane Block — Parasternal Block and Recto-Intercostal Fascial Plane Block:Superficial PSB is performed bilaterally with the patient in the supine position using a high-frequency linear USG probe. The probe is inserted longitudinally 2cm lateral to the sternal border to visualize the T2T4 intercostal space and identify the pectoralis major muscle, intercostal muscle, and pleura. Using an in-plane approach with a 100mm needle, 10ml of 0.25% bupivacaine is administered between the pectoralis major and intercostal muscle. Additionally, a Recto-Intercostal Fascial Plane Block is performed bilaterally with a high-frequency linear USG probe. The probe is inserted 2-3cm lateral to the xiphoid to visualize the rectus abdominis muscle and the 6th-7th cartilages. The needle is advanced to the plane between the costal cartilage and the rectus abdominis muscle using the in-plane technique, and 1-2ml of saline is injected. After spreading to the target plane is observed, 20ml of 0.25% bupivacaine is administered.
  Arms: Parasternal Block and Recto-İntercostal Fascial Plane Block
Other: Parasternal Block and Erector Spinae Plane Block — Superficial PSB is performed with the patient in the supine position using a high-frequency linear USG probe. The probe is placed longitudinally 2cm lateral to the sternal border to identify the T2T4 intercostal space, pectoralis major muscle, intercostal muscle, and pleura. Using an in-plane approach with a 100mm needle, 10ml of 0.25% bupivacaine is applied between the pectoralis major and intercostal muscle. Additionally, an erector spinae plane block is performed with a high-frequency USG probe. Erector spinae plane block is performed under general anesthesia, in the lateral position, under USG guidance, after sterilization, by inserting a needle between the deep surface of the erector spinae muscle and the transverse process with an in-plane approach in the craniocaudal direction. If no air or blood is seen in the aspiration, a 2mL serum test dose is applied to this area and a total of 20mL of 0.25% bupivacaine is injected bilaterally to perform an erector spinae plane block.
  Arms: Parasternal Block and Erector Spinae Plane Block

SUMMARY:
The goal of this study is to compare the analgesic efficacy of the combination of PSB and RIFPB and the combination of PSB and ESPB in patients undergoing cardiac surgery with sternotomy.

DETAILED DESCRIPTION:
This study will consist of two randomized groups: Group RIFPB (n=12), Group ESP (n=12). All patients will receive standard general anesthesia. Group RIFPB patients will receive PSB and RIFPB with 0.25% bupivacaine (total volume 60 ml) bilaterally. Group ESPB patients will receive PSB and ESPB with 0.25% bupivacaine (total volume 60 ml) bilaterally. All blocks will be performed after induction of general anesthesia and before surgical incision. All patients in the study will be given 50 mg dexketoprofen and 1 g paracetamol intravenously (i.v.) 10 minutes before skin closure. Within the first 24 hours after surgery, all patients will be given 3x1 g iv paracetamol and 2x50 mg dexketoprofen. Numerical Rating Scale (NRS) will be used to assess postoperative pain at 1, 6, 12, 18 and 24 hours. All patients will receive morphine via a patient-controlled analgesia (PCA) device within 24 hours of surgery. If pain score is ≥ 4 despite this protocol, 50 mg tramadol iv (maximum dose 300 mg/day) will be administered as rescue analgesia.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients over 18 years of age who will undergo cardiac surgery with sternotomy under general anesthesia and who are in classes I-IIIII according to the American Society of Anesthesiologists (ASA) risk classification.

Exclusion Criteria:

* Patients who did not give consent,
* patients with coagulopathy,
* patients with signs of infection at the block application site,
* patients using anticoagulants,
* patients with local anesthetic drug allergies,
* patients with unstable hemodynamics,
* patients who could not cooperate during postoperative pain assessment

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-08-15 (Estimated); Primary Completion 2024-09-15 (Estimated); Study Completion 2024-09-20 (Estimated)

PRIMARY OUTCOMES:
Comparing the numerical rating scale scores | Postoperative 24 hours
  Numerical rating scale will be used for pain assessment. The scores of the numerical rating scale changes between 0 to 10 points. 10 points mean "the most severe pain that the patient ever had". 0 point means "there is no pain." Higher scores mean worse outcome.

SECONDARY OUTCOMES:
Comparing total morphine consumption | Postoperative 24 hours
  Postoperative analgesic need

CONTACTS AND LOCATIONS:
Overall Officials: Oğuz Gündoğdu, Principal Investigator — Sivas Cumhuriyet University School of Medicine, Anesthesiology and Reanimation